CLINICAL TRIAL: NCT01419340
Title: An Open Label, Randomized, 2-Period, 2-Treatment, Crossover, Single-Dose Bioequivalence Study of Donepezil Hydrochloride Tablets 10mg [Test Formulation, Torrent Pharmaceutical Limited., India] Versus Aricept® (Donepezil Hydrochloride) Tablets 10mg [Reference Formulation, Eisai Inc.), in Healthy Human Volunteers Under Fasting Conditions.
Brief Title: Bioequivalence Study of Torrent Pharmaceutical Limited's Donepezil Hydrochloride Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Chief Investigator, Torrent Pharmaceuticals Limited
Other Study IDs: PK-07-116
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Healthy

INTERVENTIONS:
Drug: Torrent's Donepezil Hydrochloride Tablets 10mg

SUMMARY:
Objective:

To compare the rate and extent of release of the drug substance from the two tablet formulation of Donepezil Hydrochloride Tablets 10mg of Torrent Pharmaceuticals Limited and the Aricept® Tablets 10mg of Eisai Inc., Dosing periods were separated by a washout period of at least 7 days.

Study Design:

Randomized, open label, two treatment, two period, two sequence, single dose, crossover study in healthy human adult subjects

ELIGIBILITY:
Inclusion Criteria:

* The volunteers were excluded from the study based on the following criteria:

  * Sex: male.
  * Age: 18 - 45 years. .
  * Volunteer with BMI of 18-27 (inclusive both) kg/m2 with minimum of 50 kg weight.
  * Healthy and willing to participate in the study.
  * Volunteer willing to adhere to the protocol requirements and to provide written informed consent.
  * Non-smokers or smoker who smokes less than 10 cigarettes per day

Exclusion Criteria:

* The volunteers were excluded from the study based on the following criteria:

  * Clinically relevant abnormalities in the results of the laboratory screening evaluation.
  * Clinically significant abnormal ECG or Chest X-ray.
  * Systolic blood pressure less than 100 mm Hg or more than 140 mm Hg and diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
  * Pulse rate less than 50/minute or more than 100/minute.
  * Oral temperature less than 95°P or more than 98.6°P.
  * Respiratory rate less than 12/minute or more than 20/minute
  * History of allergy to the test drug or any drug chemically similar to the drug under investigation.
  * History of alcohol or drug abuse
  * Positive breath alcohol test
  * Recent history of kidney or liver dysfunction.
  * History of consumption of prescribed medication since last 14 days or OTC medication since last 07 days before beginning of the study.
  * Volunteers suffering from any chronic illness such as arthritis, asthma etc.
  * History of heart failure.
  * HIV, HCV, HBsAg positive volunteers.
  * Opiate, tetra hydrocannabinol, amphetamine, barbiturates, benzodiazepines, - - Cocaine positive volunteers based on urine test.
  * Volunteers suffering from any psychiatric (acute or chronic) illness requiring medications.
  * Administration of any study drug in the period 0 to 3 months before entry to the study.
  * History of significant blood loss due to any reason, including blood donation in the past 3 months.
  * History of pre-existing bleeding disorder.
  * Existence of any surgical or medical condition, which, in the judgment of the chief investigator and/or clinical investigator/physician, might interfere with the absorption, distribution, metabolism or excretion of the drug or likely to compromise the safety of volunteers.
  * Inability to communicate or co-operate due to language problem, poor mental development or impaired cerebral function.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult

PRIMARY OUTCOMES:
bioequivalence based on Composite of Pharmacokinetics
  bioequivalence; 90% geometric confidence interval of the ratio of least-squares means of the test to reference product should be within 80.00% - 125.00% for AUC-unf, AUCo-t and Cmax.

CONTACTS AND LOCATIONS:
Locations (1):
- Bio Evaluation Centre, Torrent Pharmaceuticals Ltd.,, Village Bhat, Gandhinagar, Gujarat, India